CLINICAL TRIAL: NCT03948243
Title: Licorice Botanical Dietary Supplements - Metabolism and Safety in Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Oregon State University (Other)
Responsible Party: Principal Investigator, Richard B van Breemen, Professor, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019-0115
Record Dates: First submitted 2019-05-08; First posted 2019-05-13 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Food-drug Interaction
Keywords: Licorice
MeSH Terms: interventions — Glycyrrhiza glabra extract; Alprazolam; Caffeine; Tolbutamide; Dextromethorphan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- G.Glabra (Experimental): single arm
  Interventions: Dietary Supplement: Licorice; Drug: Alprazolam 2 MG; Drug: Caffeine 100 MG; Drug: Tolbutamide 250 mg; Drug: Dextromethorphan 30mg

INTERVENTIONS:
Dietary Supplement: Licorice — Experimental :G. glabra Licorice extract: 2 gelatin capsules (75 mg) per day for 14 days
  Other Names: G. glabra
Drug: Alprazolam 2 MG — probe substrate
  Other Names: CYP3A4/5 substrate
Drug: Caffeine 100 MG — probe substrate
  Other Names: CYP1A2 substrate
Drug: Tolbutamide 250 mg — probe substrate
  Other Names: CYP2C9 substrate
Drug: Dextromethorphan 30mg — probe substrate
  Other Names: CYP2D6 substrate

SUMMARY:
Human safety studies will be carried out to test whether red clover botanical dietary supplements used by peri- and post-menopausal women are safe to use with Food and Drug Administration (FDA)-approved drugs. To test this, a red clover dietary supplement (previously tested in women at the University of Illinois at Chicago without any harmful effects) will be given with four selected FDA-approved drugs to determine if the Licorice supplement can increase or decrease how these medications are absorbed, metabolized and excreted by the human body. Preclinical studies predict that the licorice supplement might affect the metabolism or break down of these probe drugs.

DETAILED DESCRIPTION:
At the start of a study, subjects will be administered low doses of a mixture of four FDA-approved drugs (caffeine, tolbutamide, dextromethorphan, and alprazolam), and serial blood samples will be drawn and analyzed for the concentration of each drug over time. Afterwards, participants will take the licorice dietary supplement twice daily for 14 days to allow for potential inhibition or induction of drug metabolizing enzymes and transporters. Thereafter, the same drugs will be taken again to obtain a second measure of drug concentrations in blood over time. Changes in the concentration-time curve values for each probe drug obtained before and after ingestion of the supplement would indicate that metabolism of the probe drugs is impacted by the licorice dietary supplement.

ELIGIBILITY:
Inclusion Criteria:

* healthy peri- and post-menopausal women ages 40 - 79
* non-smokers
* no-significant medical conditions as assessed by subject-reported medical history, physical examination and blood and urine chemistry screens
* no medical condition that requires chronic use of medication

Exclusion Criteria:

* known allergies or hypersensitivity to caffeine, dextromethorphan, sulfonylureas (tolbutamide), benzodiazepines, or licorice
* positive pregnancy test
* use of hormone therapy within 8 weeks of study initiation for oral agents, 4 weeks for transdermal or other topical agents
* use of caffeine products 7 days before study participation or during the study
* use of citrus products 7 days before study participation or during the study
* other prescription (with the exception of the Mirena® IUD) or non-prescription medicines within the 2 weeks prior to study initiation or during the study
* chronic diseases, such as inflammatory bowel disease, that could alter the absorption or metabolism of the probe substrates
* unwillingness to comply with study requirements
* current participation in another clinical trial
* CYP2D6 deficiency based on phenotyping at screening
* smoker
* licorice (whether as a botanical dietary supplement, candy, food, drink or otherwise) within the previous two weeks and during the study
* use of any dietary supplements within the last 2 weeks prior to study initiation and during the study
* extreme obesity (defined as >40 BMI)
* alcohol or drug abuse
* chronic diseases such as diabetes.

Ages: 40 Years to 79 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 19 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2022-04-22 (Actual)

PRIMARY OUTCOMES:
1. Area Under the Curve (AUC) | baseline and 14 days
  Concentration of probe drugs from blood draws during the 14-day intervention will be used to calculate area under the (extrapolated) concentration-time curve to determine any changes compared to pre-intervention.

SECONDARY OUTCOMES:
1. Apparent Clearance | baseline and 14 days
  Concentration of probe drugs from blood draws during the 14-day intervention will be used to calculate apparent clearance of probe drug to determine any changes compared to pre-intervention.
2. Peak Concentration | baseline and 14 days
  Concentration of probe drugs from blood draws during the 14-day intervention will be used to calculate peak concentration of probe drug to determine any changes compared to pre-intervention.
3. Time for Peak Concentration | baseline and 14 days
  Concentration of probe drugs from blood draws during the 14-day intervention will be used to calculate time for peak concentration of probe drug to determine any changes compared to pre-intervention.
4. Drug Half-life [Time Frame: baseline and 14 days] | baseline and 14 days
  Concentration of probe drugs from blood draws during the 14-day intervention will be used to calculate half-life of probe drug to determine any changes compared to pre-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Richard vanBreemen, PhD, Study Director — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No